CLINICAL TRIAL: NCT02173951
Title: A Decisional Algorithm to Start Iron Chelation in Minimally Transfused Young Beta-thalassemia Major Patients Naive to Iron Chelation Therapy. A Comparative Randomized Prospective Study
Brief Title: An Algorithm to Start Iron Chelation in Minimally Transfused Young Beta-thalassemia Major Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, Professor of pediatric, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: start of ICT in young BTM
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Beta Thalassemia Major
Keywords: young minimally transfused beta thalassemia major; labile plasma iron (LPI); Transferrin saturation (TSAT); Deferiprone; Transfusional iron loading rate; Transfusion units
MeSH Terms: conditions — beta-Thalassemia | interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm 1 iron chelation (Active Comparator): Active Comparator arm : iron chelation Included 32 thalassemia major patients with low serum ferritin (≥500) . They will receive low dose Deferiprone( DFP )on 50 mg/kg/d.
  Interventions: Drug: Deferiprone
- arm 2 blood transfusion (Placebo Comparator): Placebo Comparator arm: blood transfusion only Included 32 thalassemia patients with low serum ferritin (≥500). They receive blood transfusion with no chelation. Patients will start deferiprone 75 mg/kg/d when reaching Primary end point which is elevation of SF to around 1000 ng/ml or more or Tsat > 90 % and or LPI > 0.6
  Interventions: Drug: Deferiprone

INTERVENTIONS:
Drug: Deferiprone — in arm 1 ( active comparator) will receive a starting dose of Deferiprone (DFP) 50mg⁄ kg ⁄ d, administered orally 3 times daily. Routine dose adjustments will be made according to serum ferritin trends and safety.
  Patients reaching serum ferritin ≥1000 will be subjected to dose escalation of DFP to 75 mg/kg/d.
  Patients in Placebo Comparator arm when reaching end point elevation of SF to around 1000 ng/ml or more or Tsat > 90 % and or LPI > 0.6 will start deferiprone 75 mg/kg/d
  Other Names: ferriprox

SUMMARY:
A prospective randomized study on Safety, Tolerability and Efficacy of oral Low dose DFP (50 mg/kg/day) in minimally transfused B-TM after 5 transfusions when SF reaches 500 ng/m and with either appearance of LPI > 0.2 or TSAT reaches 50% compared with non treatment arm.

So the aim of this study:

1. To determine the time as well as amount of transfused iron ( calculated in mg iron/kg ) which lead to Serum ferritin reaches 500 ng /ml and LPI appearance >0.2 as well as TSAT reaches 50 % .
2. Tolerability and safety of early low dose DFP 50mg/kg and effectiveness to postpone or prevent SF from reaching 1000 ng/ml or LPI >0.6 or TSAT >70% in comparison to patients not starting chelation therapy
3. Determine adverse events whether drug or non drug related

DETAILED DESCRIPTION:
This is a 1 year randomized prospective study that will include 64 patients with β-thalassemia major 6-36 months, those already engaged in transfusion program and received 5-7 transfusions recruited from the thalassemia clinic children hospital Ain Shams University. Consents will be taken from patient or legal guardian after explaining to them the nature of the study.

Inclusion criteria

1. Young beta thalassemia major patients (diagnosed by HPLC, CBC) who started transfusion therapy who received 5-7transfusions or less, aged more than 6 months.
2. Pre-transfusional Hb should be >9 g/dL.
3. Serum ferritin should be ≤ 500ng/ml, transferrin saturation ≤ 50%.

Exclusion criteria:

1. Beta thalassemia intermedia patients, patients with other transfusion dependent anemias (myelodysplasia, other chronic hemolytic anemias , pure red cell aplasia , aplastic anemia )
2. Patients with levels of ALT >5 the upper limit of normal (ULN), serum creatinine > ULN on 2 measurements.
3. Patients with history of agranulocytosis [absolute neutrophil count (ANC) <0.5×109/L].
4. Non complaint patients acknowledged by reviewing the patient's records.

Enrollment period: expected to be 6 months period with a mean follow up period 12 months.

Randomization: the patients enrolled as they entered the study and randomised alternatively either to arm 1 or 2 using a closed envelope system that devised by the statistician

Sample size: It was calculated to be 32 patients in each study group to detect significant difference at 0.05 with study power 95%

Arms, Groups and Cohorts:

Sixty-four thalassemia major patients naive to chelation therapy will be randomized into 2 groups: 1st group: with DFP 50 mg/kg for 12 months or 2nd group: no treatment arm

Active Comparator arm : iron chelation Included 32 thalassemia major patients with low serum ferritin (≥500) . They will receive low dose DFP on 50 mg/kg/d.

Placebo Comparator arm: blood transfusion only Included 32 thalassemia patients with low serum ferritin (≥500). They receive blood transfusion with no chelation. Primary end point is elevation of SF to around 1000 ng/ml or more or Tsat > 90 % and or LPI > 0.6 Both groups will be followed up with intervals of 3 months both clinically and laboratory with a mean time of 12 months.

Patients reaching serum ferritin ≥1000 will be subjected to dose escalation of DFP to 75 mg/kg/d.in Active Comparator arm and start of DFP 75MG/KG/D in Placebo Comparator arm.

Study procedures:

1. Medical records of thalassemia patients will be reviewed & data will be gathered including:

   * Age at onset.
   * Transfusion history:

     * Amount in each transfusion: grams of administered RBCs
     * Frequency.
     * Calculation of the transfusion index in ml packed red cell per body weight in Kg per year.
     * Transfusional iron loading rate: This will be calculated from the blood volume transfused between baseline and the end of the study. The average iron content per transfusion unit, derived from the measured hematocrit. The transfusional iron loading rate will be then expressed in mg of the transfused iron per kg body weight per day.
   * History of viral hepatitis (hepatitis B and C virus).
2. Laboratory investigations:

   1. Pre-transfusion Complete blood picture (Both manual and electronic ANC ).
   2. Liver and kidney functions.
   3. LPI, Serum Ferritin, serum iron and transferring saturation measurement :

Serum ferritin, transferring saturation (TSAT) and LPI will be checked prior to transfusion at base line, 3, 6, 9, and 12 month interval.

Positive predictive value of LPI will be estimated in relation to TSAT, SF, frequency of blood transfusion, transfusion index, and transfusional iron loading rate at which patients will start oral chelation therapy.

Compliance to ICT: Compliance to chelation therapy was assessed by reviewing patient self-report of dose-taking and the appropriate number of doses taken during each day was checked by prescription refills and measure amount of the drug in the retained bottles; a cutoff point below 70% was considered as poor compliance to the regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Young beta thalassemia major patients (diagnosed by HPLC, CBC) who started transfusion therapy who received 5-7transfusions or less, aged more than 6 months.
2. Pre-transfusional Hb should be >9 g/dL.
3. Serum ferritin should be ≤ 500ng/ml, transferrin saturation ≤ 50%.

Exclusion Criteria:

* 1. Beta thalassemia intermedia patients, patients with other transfusion dependent anemias (myelodysplasia, other chronic hemolytic anemias , pure red cell aplasia , aplastic anemia ) 2. Patients with levels of ALT >5 the upper limit of normal (ULN), serum creatinine > ULN on 2 measurements.

  3. Patients with history of agranulocytosis [absolute neutrophil count (ANC) <0.5×109/L].

  4. Non complaint patients acknowledged by reviewing the patient's records.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
determine the time and number of transfusion units as well as amount of infused iron that will lead to appearance of LPI >0.2 or TSAT>50 % , serum ferritin ≥ 500 ng/ml in the studied thalassemic patients which warrant start of iron chelation | 12 months
  To determine the time as well as amount of transfused iron ( calculated in mg iron/kg ) at which there is LPI appearance of >0.2 as well as TSAT reaching 70 %, a serum ferritin ≥ 500 in order to start Iron chelation therapy

SECONDARY OUTCOMES:
Evaluation of safety of early use of iron chelation Therapy (ICT) in terms of drug related AEs or SAEs | 12 months
  To determine the Tolerability and safety of early low dose DFP 50mg/kg and effectiveness to postpone or prevent SF from reaching 1000 ng/ml or LPI >0.6 or TSAT >70% in comparison to patients not starting chelation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen S Elalfy, professour, Principal Investigator — Ain Shams University
Locations (1):
- Pediatric Hematology clinic, Ain Shams University, Cairo, Egypt

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597
- [Derived] Elalfy MS, Adly A, Awad H, Tarif Salam M, Berdoukas V, Tricta F. Safety and efficacy of early start of iron chelation therapy with deferiprone in young children newly diagnosed with transfusion-dependent thalassemia: A randomized controlled trial. Am J Hematol. 2018 Feb;93(2):262-268. doi: 10.1002/ajh.24966. Epub 2017 Nov 27. PMID 29119631